CLINICAL TRIAL: NCT03772041
Title: A Multicenter, Double-blind, Randomized, Active-controlled, Parallel-group, Non-inferiority Trial to Evaluate the Efficacy and Safety of OPC-61815 Injection Compared With Tolvaptan 15-mg Tablet in Patients With Congestive Heart Failure
Brief Title: Efficacy and Safety Trial of OPC-61815 Injection Compared With Tolvaptan 15-mg Tablet in Patients With Congestive Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 263-102-00003; JapicCTI-184234 (Other: Japic)
Record Dates: First submitted 2018-12-05; First posted 2018-12-11 (Actual); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPC-61815 injection 16 mg (Experimental): Once daily for 5 days placebo tablet will be orally administered, followed immediately by intravenous administration of OPC-61815 at 16 mg
  Interventions: Drug: OPC-61815
- Tolvaptan tablet 15mg (Active Comparator): Once daily for 5 days tolvaptan 15-mg tablet will be orally administered, followed immediately by 1-hour intravenous administration of placebo
  Interventions: Drug: Tolvaptan Tab 15 MG

INTERVENTIONS:
Drug: OPC-61815 — Once daily for 5 days placebo tablet will be orally administered, followed immediately by intravenous administration of OPC-61815 at 16 mg
  Arms: OPC-61815 injection 16 mg
Drug: Tolvaptan Tab 15 MG — Once daily for 5 days tolvaptan 15-mg tablet will be orally administered, followed immediately by 1-hour intravenous administration of placebo
  Arms: Tolvaptan tablet 15mg

SUMMARY:
To confirm the non-inferiority of OPC-61815 16-mg injection to tolvaptan 15-mg tablet using as the primary endpoint the change in body weight following 5-day intravenous administration of OPC-61815 16-mg injection or 5-day oral administration of tolvaptan 15-mg tablet to CHF patients with volume overload despite having received diuretics other than vasopressin antagonists

ELIGIBILITY:
Inclusion Criteria:

* Patients who are currently on treatment with any of the following diuretics

  1. Loop diuretics equivalent to furosemide tablet or fine granules at a dose of 40 mg/day or higher
  2. Concomitant use of a loop diuretic and a thiazide diuretic (including thiazide analogs) at any dose
  3. Concomitant use of a loop diuretic and an aldosterone antagonist or potassium-sparing diuretic agent at any dose
* Patients with congestive heart failure in whom lower limb edema, pulmonary congestion, and/or jugular venous distension due to volume overload is present
* Patients who are currently hospitalized or who are able to be hospitalized during the trial

Exclusion Criteria:

* Patients with acute heart failure
* Patients who are on a ventricular assist device
* Patients who are unable to sense thirst or who have difficulty with fluid intake

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Sato, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Saiseikai Kumamoto Hospital, Kumamoto, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to https://clinical-trials.otsuka.com/contact-us
URL: https://clinical-trials.otsuka.com/contact-us

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OPC-61815 Injection 16 mg | Tolvaptan Tablet 15mg
Started | 149 | 145
Completed | 135 | 135
Not Completed | 14 | 10
Not completed — Adverse Event | 8 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 4 | 2
Not completed — Physician Decision | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPC-61815 Injection 16 mg | Tolvaptan Tablet 15mg | Total
Number analyzed (Participants) | 149 | 145 | 294
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.0 (10.2) | 75.4 (8.2) | 74.7 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 47 | 84
  Male | 112 | 98 | 210
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 149 | 145 | 294
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 149 | 145 | 294

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Body Weight
Description: Change in body weight from baseline (before investigational medicinal product [IMP] administration on Day 1) at time of final IMP administration (day after final IMP administration). A negative change from baseline indicates improvement.
Time Frame: Baseline, Day 6
Population: Full Analysis Set: subjects who received at least one dose of IMP and had at least one postbaseline weight measurement
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | OPC-61815 Injection 16 mg | Tolvaptan Tablet 15mg
Number analyzed (Participants) | 149 | 144
kg | -1.67 [-1.93 to -1.41] | -1.36 [-1.62 to -1.10]

2. Secondary Outcome: Improvement Rate for Lower Limb Edema and Pulmonary Congestion
Description: The improvement rate was defined as the percentage of subjects in whom the symptom was present at baseline and it markedly improved or improved after IMP administration. Improvement category is a 4-point scale below:
  * Markedly improved
  * Improved
  * Unchanged
  * Deteriorated
Time Frame: Baseline, Day 6
Population: Full Analysis Set: subjects who received at least one dose of IMP and had at least one postbaseline weight measurement were included in the full analysis. "Number Analyzed" = number of subjects with baseline symptoms.
Measure: Number; unit: percentage of participants
Arm/Group | OPC-61815 Injection 16 mg | Tolvaptan Tablet 15mg
Number analyzed (Participants) | 149 | 145
percentage of participants
  Lower Limb Edema: number analyzed (Participants) | 122 | 111
  Lower Limb Edema | 68.9 | 75.7
  Pulmonary Congestion: number analyzed (Participants) | 123 | 119
  Pulmonary Congestion | 56.1 | 64.7

3. Secondary Outcome: Change From Baseline in Jugular Venous Distension and Hepatomegaly
Description: * Jugular Venous Distension: the presence of Jugular Venous Distension was checked, and if present, the height (in cm) from the sternal angle to the highest point of pulsation in the internal Jugular vein was measured with the subject in a semi-upright position. A negative change from baseline indicates improvement.
  * Hepatomegaly: the presence of a palpable liver was checked, and if present, the width (distance from the right costal arch of the right chest, in cm) was measured. A negative change from baseline indicates improvement.
Time Frame: Baseline, Day 6
Population: Subjects with baseline values in the Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: cm
Arm/Group | OPC-61815 Injection 16 mg | Tolvaptan Tablet 15mg
Number analyzed (Participants) | 149 | 145
cm
  Jugular Venous Distension: number analyzed (Participants) | 52 | 59
  Jugular Venous Distension | -2.89 [-3.45 to -2.33] | -3.15 [-3.68 to -2.62]
  Hepatomegaly: number analyzed (Participants) | 12 | 10
  Hepatomegaly | -0.93 [-1.44 to -0.43] | -0.88 [-1.43 to -0.33]

4. Secondary Outcome: Percentage of Subjects Who Achieve Resolution of Pulmonary Rales and Third Cardiac Sound
Description: Percentage of subjects in whom the symptom was present at baseline and disappeared after IMP administration was provided.
  * The presence of pulmonary rales was checked by auscultation.
  * The presence of cardiac third sound was checked by auscultation.
Time Frame: Baseline, Day 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | OPC-61815 Injection 16 mg | Tolvaptan Tablet 15mg
Number analyzed (Participants) | 149 | 145
percentage of participants
  Pulmonary Rales: number analyzed (Participants) | 35 | 19
  Pulmonary Rales | 74.3 | 78.9
  Third Cardiac Sound: number analyzed (Participants) | 41 | 42
  Third Cardiac Sound | 31.7 | 31.0

5. Secondary Outcome: Improvement Rate for New York Heart Association (NYHA) Classification
Description: NYHA classification assesses the severity of heart failure based on subjective symptoms as follows.
  Class I: No limitations of physical activity. Ordinary physical activity caused no undue fatigue, palpitation, dyspnea or anginal pain.
  Class II: Slight limitation of physical activity, comfortable at rest. Ordinary physical activity resulted in fatigue, palpitation, dyspnea or anginal pain.
  Class III: Marked limitation of physical activity, comfortable at rest. Less than ordinary physical activity caused fatigue, palpitation, dyspnea or anginal pain.
  Class IV: Inability to carry on any physical activity without discomfort. heart failure or anginal syndrome may have been present even at rest. If any physical activity was undertaken, discomfort was increased.
  Of the subjects with Class II or higher at baseline, the percentage of subjects whose NYHA classification stage at the time of final IMP administration improved by 1 or more grades was provided.
Time Frame: Baseline, Day 6
Population: Full Analysis Set: subjects who received at least one dose of IMP and had at least one postbaseline weight measurement were included in the full analysis. "Overall Number of Participants Analyzed" = number of subjects with a baseline of class II or more.
Measure: Number; unit: percentage of participants
Arm/Group | OPC-61815 Injection 16 mg | Tolvaptan Tablet 15mg
Number analyzed (Participants) | 136 | 120
percentage of participants | 44.9 | 42.5

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from the start of IMP administration up to 15 days
Description: Subjects who received at least one dose of IMP were included in the safety analysis.
Arm/Group | OPC-61815 Injection 16 mg | Tolvaptan Tablet 15mg
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/145
Serious Adverse Events (participants affected / at risk) | 6/149 | 5/145
Other Adverse Events (participants affected / at risk) | 61/149 | 57/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-61815 Injection 16 mg (N=149) | Tolvaptan Tablet 15mg (N=145)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
General infarction (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-61815 Injection 16 mg (N=149) | Tolvaptan Tablet 15mg (N=145)
Anaemia (Blood and lymphatic system disorders) | 3 | 4
Atrial fibrillation (Cardiac disorders) | 1 | 3
Ventricular tachycardia (Cardiac disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 9 | 9
Dry mouth (Gastrointestinal disorders) | 4 | 8
Nausea (Gastrointestinal disorders) | 3 | 0
Pyrexia (General disorders) | 4 | 2
Thirst (General disorders) | 13 | 16
Blood potassium increased (Investigations) | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 15 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 3
Hypernatraemia (Metabolism and nutrition disorders) | 4 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 1
Renal impairment (Renal and urinary disorders) | 4 | 2
Eczema (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 3
Hypotension (Vascular disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT03772041/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT03772041/SAP_001.pdf